CLINICAL TRIAL: NCT01500408
Title: A Randomized, Single-Blind, Crossover Study in Healthy Volunteers to Demonstrate the Bioequivalence of Interferon Beta-1a Manufactured by Two Different Processes
Brief Title: Demonstrate the Bioequivalence of Interferon Beta-1a (INFB) Manufactured by Two Different Processes in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: 108HV106
Record Dates: First submitted 2011-12-22; First posted 2011-12-28 (Estimated); Last update posted 2012-11-19 (Estimated); Status verified 2012-11

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1a

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Commercial INFB followed by Investigational INFB (Other): Process A (currently-approved manufacturing process involving FBS) first, then Process B (new serum-free manufacturing process, without FBS)
  Interventions: Drug: Interferon beta-1a (current approved manufacturing process invloving FBS); Drug: Interferon beta-1a (new process, manufactured without FBS)
- Investigational INFB followed by Commercial INFB (Other): Process B (new serum-free manufacturing process, without FBS) first, then Process A (currently-approved manufacturing process involving FBS)
  Interventions: Drug: Interferon beta-1a (current approved manufacturing process invloving FBS); Drug: Interferon beta-1a (new process, manufactured without FBS)

INTERVENTIONS:
Drug: Interferon beta-1a (current approved manufacturing process invloving FBS) — Single dose of 60 mcg given Intramuscularly (IM)
  Other Names: Avonex®)
Drug: Interferon beta-1a (new process, manufactured without FBS) — Single dose of 60 mcg given Intramuscularly (IM)

SUMMARY:
Biogen Idec has developed a novel process to manufacture Interferon beta-1a (INFB), the active ingredient of Avonex®, that does not include fetal bovine serum (FBS). This bioequivalence study is being conducted to confirm the pharmacokinetic (PK) and pharmacodynamic (PD) comparability of Interferon beta-1a produced by the currently approved serum-containing process and Interferon beta-1a produced by the new serum-free manufacturing process.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authoriziation to use protected health information (PHI) in accordance with national and local subject privacy regulations.
2. Must be healthy males or females 18 to 45 years old, inclusive, at the time of informed consent.
3. Must have a body mass index (BMI) of 18.5 to 30.0 kg/ m2, inclusive, and a minimum body weight of 50.0 kg at Screening and Day-1 Baseline.
4. Subjects of childbearing potential must practice effective contraception during the study and be willing and able to continue contraception for 30 days after their last dose of study treatment.

Exclusion Criteria:

1. Known history of human immunodeficiency virus (HIV).
2. Positive test result at Screening for hepatitis C antibody (HCV Ab) or current hepatitis B infection (defined as positive for hepatitis surface antigen [HBcAb] at Screening). Subjects with immunity to hepatitis B from either active vaccination (defined as negative HBsAg, positive hepatitis B surface anitbody [HBsAg], and negative HBcAb) or from previous natural infection (defined as negative HBsAg, positive HBsAb immunoglobulin G, and positiveHBcAb) are eligible to participate in the study (definitions are based on the Centers for Disease Control and Prevention interpretation of the hepatitis B serology panel).
3. Subjects with a history of malignant disease, including solid tumors and hematologic malignancies (except basal cell and squamos cell carcinomas of the skin that have been completely excised and are considered cured).
4. History of severe allergic or anaphylactic reactions.
5. Known allergy to any component of the IFN B-1a formulation, including a dry rubber allergy.
6. History of any clinically significant cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, or other major disease, as determined by the Investigator.
7. History of seizure disorder or unexplained blackouts.
8. History of suicidal ideation or an episode of clinically severe depression (as determined by the Investigator).
9. Serious local infection (e.g., cellulitis, abscess) or systemic infection (pneumonia, septicemia), at the discretion of the Investigator, within 3 months prior to Day 1.
10. History of drug or alcohol abuse (as defined by the Investigator) within 6 months prior to Screening.
11. Positive testing for drugs and alcohol at Screening or baseline (Day-1).
12. Alcohol use within 48 hours prior to Day 1. Subjects must be willing to restrict alcohol use throughout their participation in the study. Subjects may not consume more than 1 alcoholic beverage per day during this study where 1 alcoholic beverage is defined as ≤8 ounces of beer or ≤4 ounces of wine.
13. Fever (body temperature >38°C) or symptomatic viral or bacterial infection (including upper respiratory infection) within 1 week prior to Day 1.
14. Clinically significant abnormal clinical laboratory test values, as determined by the Investigator, or any values for alanine aminotransferase (ALT), aspartate aminotransferase (AST), or creatinine that are above the upper limit of normal, any values for platelets or hemoglobin that are below the lower limit of normal, or any out of normal range values for white blood cells, serum sodium, or serum potassium.
15. Any previous treatment with any interferon product, including investigational use.
16. History of hypersensitivity or intolerance to acetaminophen (paracetamol), ibuprofen, naproxen, or aspirin that would preclude use of at least 1 of these during the study.
17. Prior treatment with any investigational drug within the 30 days prior to Day 1, or within 5 half-lives of the drug, whichever is longer.
18. Treatment with any medication including over-the-counter (OTC) products within 48 hours prior to Day 1, except for the following treatments, which are allowed: contraceptives, hormone replacement therapy (HRT), local, non-systemically absorbed steroids (i.e., topical, nasal/inhaled), acetaminophen (paracetamol), ibuprofen, naproxen, and/or aspirin.
19. Female subjects who are pregnant or currently breastfeeding or have a positive pregnancy test result.
20. Vaccinations within 4 weeks prior to Day 1.
21. Blood donation (1 unit or more) within 1 month prior to Day 1.
22. Current enrollment in any other study treatment or disease study.
23. Inability to comply with study requirements.
24. Other unspecified reasons that, in the opinion of the Investigator or Biogen Idec, make the subject unsuitable for enrollment.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2012-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Area under the serum concentration-time curve (AUC) as a measure of PK. | Subjects will be followed for the duration of the study, 22 days. PK samples will be taken 5 to 60 minutes prior to dosing, and post dose at hours 2, 4, 6, 9, 12, 15, 18, 21, 24, 30, 36, 48, 72, 96 and 168.

SECONDARY OUTCOMES:
The observed maximum (peak) serum Interferon beta-1a concentration (Cmax) | Subjects will be followed for the duration of the study, 22 days. PK samples will be taken 5 to 60 minutes prior to dosing, and post dose at hours 2, 4, 6, 9, 12, 15, 18, 21, 24, 30, 36, 48, 72, 96 and 168.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Saint Paul, Minnesota, United States